CLINICAL TRIAL: NCT05037045
Title: Department of Pharmacy, the Affiliated Hospital of Xuzhou Medical University
Brief Title: Effect of Gene Polymorphisms on GLP-1 Receptor Agonists Response in Patients With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2018-KL085
Record Dates: First submitted 2021-08-27; First posted 2021-09-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2DM; GLP-1 RA; gene polymorphism
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLP-1 RA therapy (Experimental): GLP-1 RA was injected subcutaneously at standard dose and frequency for consecutive 6 months.
  Interventions: Drug: GLP-1 receptor agonist

INTERVENTIONS:
Drug: GLP-1 receptor agonist — GLP-1 RA was injected subcutaneously at standard dose and frequency for consecutive 6 months in patients with T2DM
  Other Names: GLP-1 analogues

SUMMARY:
1. This is an prospective study to evaluate the effect of gene polymorphisms on therapeutic responses to glucagon like peptide-1 receptor agonist (GLP-1 RA) in patients with T2DM.
2. T2DM patients and healthy subjects were recruited to identify genotypes and detect the level of T2DM susceptibility genes expression levels in the plasma of healthy participants and T2DM patients.
3. This is a retrospective cohort study of patients with T2DM who were treated with exenatide twice daily as a part of their diabetes care for at least 12 months.

DETAILED DESCRIPTION:
Many guidelines recommend the preferential use of GLP-1 RA after single drug or multiple oral hypoglycemic drugs and basic insulin therapy for poor glycemic control. However, the clinical responsiveness to GLP-1 RA varies among patients with T2DM. It has been reported that genetic factors are the important reasons for individual variation in therapeutic response of antidiabetic drugs. At present, dozens of gene loci related to therapeutic response of antidiabetic drugs have been screened, which are of great clinical significance in guiding clinical individualized treatment, improving the efficacy and safety of drugs, and reducing the drug costs.

GLP-1 RA was injected subcutaneously at standard dose and frequency for consecutive 6 months. The patients were visited at moths 0, 3, and 6, and medical histories, physical examinations, and routine clinical laboratory tests were performed during these visits. The general anthropometric parameters considered for this study were height (m), weight (kg), and waist and hip circumferences (cm) at baseline, 3 months and 6months after exenatide treatment. After an overnight fast, venous blood samples were obtained both in the fasting state and 2 h later during a standard 75-g oral glucose tolerance test. Parameters were measured at baseline, the end of months 3 and 6 after administration of exenatide.

Peripheral blood was collected at follow-up and genomic DNA was extracted from peripheral blood leucocytes. We further explored the association of gene polymorphisms with the therapeutic effect of GLP-1 RA in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of T2DM；
2. a body mass index (BMI) of 20-35 kg/m2；
3. an HbA1c of 7.0%-12%, an age of 25-70 years；
4. required data available at baseline, 3 months, and 6 months after GLP-1 RA therapy.

Exclusion Criteria:

1. Patients with serious diseases such as acute myocardial infarction, cerebral vascular accident, trauma, kidney or liver diseases, severe gastrointestinal dysfunction, and history of pancreatitis；
2. patients receiving GLP-1 analogues, weight loss drugs, glucocorticoids, drugs affecting gastrointestinal peristalsis in the past 3 months；
3. those with missing data at the time points of baseline, 3 months, and 6 months after GLP-1 RA therapy.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline HbA1c at 1 month | 1 month after GLP-1 RA treatment
  In order to observe the change from baseline HbA1c at 1 month after GLP-1 RA treatment
Change from baseline FPG at 1 month | 1 month after GLP-1 RA treatment
  In order to observe the change from baseline FPG at 1 month after GLP-1 RA treatment
Change from baseline PPG at 1 month | 1 month after GLP-1 RA treatment
  In order to observe the change from baseline PPG at 1 month after GLP-1 RA treatment
Change from baseline serum lipids at 1 month | 1 month after GLP-1 RA treatment
  In order to observe the change from baseline serum lipids at 1 month after GLP-1 RA treatment
Change from baseline HbA1c at 3 month | 3 month after GLP-1 RA treatment
  In order to observe the change from baseline HbA1c at 3 month after GLP-1 RA treatment
Change from baseline FPG at 3 month | 3 month after GLP-1 RA treatment
  In order to observe the change from baseline FPG at 3 month after GLP-1 RA treatment
Change from baseline PPG at 3 month | 3 month after GLP-1 RA treatment
  In order to observe the change from baseline PPG at 3 month after GLP-1 RA treatment
Change from baseline serum lipids at 3 month | 3 month after GLP-1 RA treatment
  In order to observe the change from baseline serum lipids at 3 month after GLP-1 RA treatment
Change from baseline HbA1c at 6 month | 6 month after GLP-1 RA treatment
  In order to observe the change from baseline HbA1c at 6 month after GLP-1 RA treatment
Change from baseline FPG at 6 month | 6 month after GLP-1 RA treatment
  In order to observe the change from baseline FPG at 6 month after GLP-1 RA treatment
Change from baseline PPG at 6 month | 6 month after GLP-1 RA treatment
  In order to observe the change from baseline PPG at 6 month after GLP-1 RA treatment
Change from baseline serum lipids at 6 month | 6 month after GLP-1 RA treatment
  In order to observe the change from baseline serum lipids at 6 month after GLP-1 RA treatment

SECONDARY OUTCOMES:
incidence and severity of possible adverse reaction within 1 month after GLP-1 RA treatment | 1 month after GLP-1 RA treatment
  To evaluate the incidence and severity of possible adverse reaction within 1 month after GLP-1 RA treatment, including gastrointestinal reaction and hypoglycemia
incidence and severity of possible adverse reaction within 3 month after GLP-1 RA treatment | 3 month after GLP-1 RA treatment
  To evaluate the incidence and severity of possible adverse reaction within 3 month after GLP-1 RA treatment, including gastrointestinal reaction and hypoglycemia
incidence and severity of possible adverse reaction within 6 month after GLP-1 RA treatment | 6 month after GLP-1 RA treatment
  To evaluate the incidence and severity of possible adverse reaction within 6 month after GLP-1 RA treatment, including gastrointestinal reaction and hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Renhao Wang, Ph.D, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- Department of Endocrinology, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No